CLINICAL TRIAL: NCT05787210
Title: Effects of Quadriceps Strength Training on Gait Parameters and Energy Expenditure in Children With Spastic Cerebral Palsy
Brief Title: Quadriceps Strength Training on Gait Parameters and Energy Expenditure in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0704
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Conventiional Physiotherapy
- Strength (Experimental)
  Interventions: Other: Conventiional Physiotherapy; Other: Quadriceps Strength Training

INTERVENTIONS:
Other: Conventiional Physiotherapy — The Control group will be administered with Conventional Physiotherapy that Includes 5 minutes of trunk control training, 5 minutes walking in the hall with And without the therapist assistance, walker or crutches, and finally 5 minutes of Breathing exercises for Relaxation
Other: Quadriceps Strength Training — The experimental group will be administered with the same baseline treatment such as 5 minutes of trunk control training, 5 minutes walking in the hall with or without the therapist assistance, walker or crutches and 5 minutes breathing exercises for relaxation. In addition, they were given strength training protocol intervention other than the baseline treatment. This strength training protocol include progressive resistance training program in which we gave leg lift (knee flexion and extension), Hip rotations, seated marching and the quadriceps muscles would be specifically targeted.
  Arms: Strength

SUMMARY:
The incidence of cerebral palsy is approximately 2 to 3 cases per 1000 live births around the world. In Cerebral palsy the lesion in the central nervous system frequently results in spasticity of various muscle groups. Spasticity is defined as a velocity dependent resistance to stretch. Spastic Cerebral palsy is caused by damage to the pyramidal parts of the brain.

The children with spastic CP frequently experience problems with motor control, and balance which may lead to gait abnormalities. Because of motor weakness and poor voluntary motor control the children with spastic cerebral palsy develop crouch gait characterized by excessive hip and knee flexion and a slower walking speed, a shorter stride length, and more time spent in double support. This study will help in the quality of life in spastic cerebral palsy children. This will be a Randomized Controlled Trial. Approval will be gained from the Ethical committee of the Riphah international university Lahore, Pakistan prior to the commencement of study. Written informed consent will be taken from all the patients and all information and data will be confidential. Subjects will be informed that there is no risk of study and they will be free to withdraw any time during process of study. 22 Children with Spastic CP will be randomly distributed into 2 groups. The Control Group (n=10) will be administered with the baseline treatment that Includes 5 minutes of trunk control training, 5 minutes walking in the hall with And without the therapist assistance, walker or crutches, and finally 5 minutes of Breathing exercises for Relaxation 3 sessions per week for 8 weeks. The experimental group (n=10) will be administered with the strength training intervention along with baseline treatment, 3 sessions per week for 8 weeks. Gait parameters will be evaluated physically by measuring stride and step length and cadence.

5-meter stretch test for gait parameters. the energy expenditure will be calculated by measuring the physiological cost index that includes measuring the speed of walking and resulting increase in heart rate. Data will be analyzed by using SPSS version 26.0 and necessary analysis will be done after checking the normality of Data.

ELIGIBILITY:
Inclusion Criteria:

* Diplegic Cerebral palsy
* (GMFC) level 1 and 2
* Able to follow verbal direction for standard testing

Exclusion Criteria:

* Orthopedic and Neurosurgery in last 12 months
* Children with any associated medical condition
* Children with Botox therapy in last six months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Gait parameters | Baseline and 8th week
  5-meter stretch test for gait parameters that include: the participant to walk barefoot with their normal speed on a 5-mt stretch of plain white paper with inked foot within a fixed time and it was recorded using a stopwatch. Prior to data collection, all participants had an opportunity to practice walking, as first few steps were discarded. The gait parameters analyzed will be step length, stride length, cadence and gait speed
Change in ENERGY EXPENDITURE | Baseline and 8th week
  The Physiological Cost Index was introduced by MacGregor and is used to check energy expenditure. it is calculated by estimating the speed of walking and the increase in heart rate after the child has walked a specified distance at a self-selected pace. .We calculate the physiological cost index by Formula for calculation PCI is: PCI (beats/min) = Walking heart rate
  - Resting heart rate / walking speed (m/min)

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Al-noor Special Children School, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valadao P, Piitulainen H, Haapala EA, Parviainen T, Avela J, Finni T. Exercise intervention protocol in children and young adults with cerebral palsy: the effects of strength, flexibility and gait training on physical performance, neuromuscular mechanisms and cardiometabolic risk factors (EXECP). BMC Sports Sci Med Rehabil. 2021 Feb 26;13(1):17. doi: 10.1186/s13102-021-00242-y. PMID 33637124
- [Background] Bhilwade1 DAH, DSSGP. Effect of Spasticity on Gait Parameters and Physiological Cost Index in Patients with Spastic Cerebral Palsy. 2020
- [Background] Merino-Andres J, Garcia de Mateos-Lopez A, Damiano DL, Sanchez-Sierra A. Effect of muscle strength training in children and adolescents with spastic cerebral palsy: A systematic review and meta-analysis. Clin Rehabil. 2022 Jan;36(1):4-14. doi: 10.1177/02692155211040199. Epub 2021 Aug 18. PMID 34407619